CLINICAL TRIAL: NCT06974071
Title: Effectiveness of Nonpharmacologic Therapies on Pain After Removal of Chest Drains in Postoperative Cardiac Surgery, Study Protocol
Brief Title: Effectiveness of Nonpharmacologic Therapies on Pain After Removal of Chest Drains in Postoperative Cardiac Surgery
Acronym: NPT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de La Frontera (Other)
Responsible Party: Principal Investigator, Greys Kasandra Kasandra González González, Msc., Universidad de La Frontera
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: DIM24-0009; DIM24-0009 (Other Grant/Funding Number: UNIVERSIDAD DE LA FRONTERA.)
Record Dates: First submitted 2025-05-07; First posted 2025-05-15 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Pain Management
Keywords: cardiac surgery; pain management; chest drain; non-pharmacological therapy
MeSH Terms: conditions — Agnosia | interventions — lavender oil

STUDY DESIGN:
Intervention Model Description: * Specific treatment protocol for each group. The procedures will be performed by two nurses who are part of the research, as co-investigators and project assistants, being clinical nurses of the Unit, the procedures to be performed will be assisted by Senior Nursing Technicians (TENS) on duty. This will be performed between 11:00 - 13:00, at a time to be agreed upon by the nurses, this time is preferred because of the time difference with the administration of usual analgesic treatment. The nurses do not need separate training in drain removal due to experience in the area, and the recent refresher course in the management of chest drains, and the drain removal protocol in which they participated as authors.
  * Usual treatment: Patients with indication for drainage removal after cardiac surgery, with analgesia according to the protocol indicated by the resident physician, the routine technique will be performed.
  * Experimental treatment with
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Local cold application group (Experimental): patients with indication for removal of drains after cardiac surgery, with analgesia according to the protocol indicated by the resident physician, to whom local cold will be applied . If after the removal of drains there is pain that does not subside with complementary therapy, extra analgesia may be requested.
  Interventions: Other: Local cold therapy.
- Aromatherapy group (Experimental): Patients with indication for removal of drains after cardiac surgery, with analgesia according to protocol indicated by resident physician, who at the time of removal of drains will be applied aromatherapy with lavender oil. If after the removal of drains has a pain that does not subside, with complementary therapy, you can request extra analgesia.
  Interventions: Other: Lavender oil.
- Control group. (No Intervention): Patients with indication for removal of drains after cardiac surgery, with analgesia according to the protocol indicated by the resident physician, the routine technique will be performed.

INTERVENTIONS:
Other: Local cold therapy. — It will be applied by means of a refrigerated unit based on gel pack, these units will be stored in the refrigerator of the Unit, which is kept between 2 - 6 degrees, the application protocol is described in Annex B, this was reviewed in conjunction with quality nurses of the Cardiovascular Unit, to avoid biases.
  Arms: Local cold application group
Other: Lavender oil. — Lavender essential oil will be used by applying 5 drops in a sterile dressing 15x15 which will be placed on the side of the patient's bedside at 10 cm from the patient.
  To maintain the safety of the patients and ensure the quality of the products, two essential oils will be chosen, certified by the Institute of Public Health (ISP), the first one "Lavender essential oil, body and aromatherapy use" of the Weleda brand, with sanitary authorization N° 154C-15 and the essential oil Doterra, sanitary authorization N° 2832C-6/21, with authorization by the Food and Drugs Administration (FDA), in charge of ensuring the quality of substances that are marketed from the United States to the rest of the world.
  These oils will be subjected to a characterization process, choosing the one with the highest quality and purity, through the protocol sent by the Scientific and Technological Nucleus in Bioresources (BioRen), which are specified in section 5.10.
  Arms: Aromatherapy group

SUMMARY:
The objective of this clinical trial is to determine the effectiveness of pain reduction between an experimental treatment and the usual one when removing thoracic drains in post cardiac surgery patients, in a Cardiovascular Critical Patient Unit, in Temuco, between the years 2024- 2026. Its safety will also be analyzed. The main questions to be answered are:

- What is the effectiveness of non-pharmacological therapies in reducing pain in the removal of chest drains in post-operated patient of cardiac surgery, in Cardiovascular Critical Patient Unit, Temuco, between the years 2024- 2026?

Participants:

* Two non-pharmacological therapies will be applied, to one group aromatherapy with lavender essential oils, which were previously submitted to oil property analysis. And another group with local cold therapy, there will also be a control group with the usual pharmacological therapy.
* All the groups will receive the usual pharmacological treatment, the non pharmacological therapies will only be of support, in no case they will replace the usual medical therapy.

DETAILED DESCRIPTION:
Controlled clinical trial, randomized, single-blind, with a sample of 100 postoperative cardiac surgery patients who meet inclusion and exclusion criteria. The sample will be obtained by two nurses with more than 8 years of experience in cardiac intensive care and specializations, of these patients all will receive the usual pharmacological therapy, will be divided into three groups: 25 patients (local cold); 25 patients (aromatherapy); 50 patients (with usual pharmacological therapy, indicated by medical team, without adding TNF). Data will be collected through a form. The database will be exported to STATA CORP18 software, where they will be analyzed. The ethical requirements of Ezequiel Emanuel will be considered.

Translated with DeepL.com (free version)

ELIGIBILITY:
Inclusion Criteria:

* Postoperative cardiac surgery patient with indication of the cardiac surgeon to remove chest drains within the first 24 hours postoperatively.
* Patient who follows orders and with vigil state of consciousness, temporally and spatially oriented.
* Usual analgesic treatment indicated by physician: paracetamol 1 g every 8 hours; or Metamizole 1 g every 8 hours; Ketoprofen every 8 hours, or pregabalin 75 mg every 24 hours, last administration at 07:00 am.
* INR < 2.5; Platelets > 50,000.

Exclusion Criteria:

* Patient with psychomotor agitation
* Dependence on psychotropic drugs, alcohol, or with abstinence syndrome.
* Patient in postoperative course with cardiogenic shock, with need for 2 or more vasoactive drugs (VAD).
* Older than 80 years old.
* Maintained with continuous infusion pump (CIB) of analgesia.
* Refractory pain, with second line management: Lidocaine patches, Buprenorphine patches, Patient controlled analgesia pump.
* Administration of anticoagulant at 07:00 am.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-04-20 (Actual); Primary Completion 2025-09-20 (Estimated); Study Completion 2025-12-20 (Estimated)

PRIMARY OUTCOMES:
Measurement of patient-reported pain using the visual numerical pain scale. | Pain measurement at 5, 10 and 20 minutes after drain removal.
  Pain measurement at 5, 10 and 20 minutes after drain removal. For quantification of pain using the visual numerical pain scale. it was divided into mild 1 -3 , moderate 4-6 and severe 7-10. It is necessary for the patient to understand the meaning and content of the scale, for which reason the patient must be in adequate cognitive condition to guarantee his or her ability to collaborate.

CONTACTS AND LOCATIONS:
Locations (1):
- Claro Solar 115, Temuco, Temuco, Araucanía (IX), Chile

IPD SHARING:
Plan to Share IPD: Yes
Under no circumstances will personal information of the enrolled subjects be shared, data such as:
  * Ages.
  * Pain assessment.
  * Gender.
  * Type of surgery.
  * Number of drains.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Beginning 3 months and ending 3 years after the publication of results